CLINICAL TRIAL: NCT04091451
Title: A Phase III, Randomized, Observer-blind, Placebo Controlled, Multicenter Clinical Trial to Assess Herpes Zoster Recurrence and the Reactogenicity, Safety and Immunogenicity of GSK Biologicals' Herpes Zoster Vaccine (HZ/su) When Administered Intramuscularly on a 0 and 2 Month Schedule to Adults ≥50 Years of Age With a Prior Episode of Herpes Zoster
Brief Title: Safety and Immunogenicity Study of GlaxoSmithKline's Herpes Zoster Subunit Vaccine (HZ/su) When Given on a Two-dose Schedule to Adults at Least 50 Years of Age (YOA) With a Prior Episode of Herpes Zoster
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 204939; 2016-000744-34 (EudraCT Number)
Record Dates: First submitted 2019-09-03; First posted 2019-09-16 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Herpes Zoster
Keywords: Shingles; Shingles recurrence; HZ; Vaccine response rate
MeSH Terms: conditions — Herpes Zoster | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HZ/su Group (Experimental): Participants with a prior episode of HZ randomized to the HZ/su group were scheduled to receive 2 doses of HZ/su vaccine, one at Day 1 and one at Month 2.
  Interventions: Biological: Herpes Zoster subunit (HZ/su) vaccine (GSK1437173A)
- Placebo Group (Placebo Comparator): Participants with a prior episode of HZ randomized to the Placebo group were scheduled to receive 2 doses of placebo, one at Day 1 and one at Month 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Herpes Zoster subunit (HZ/su) vaccine (GSK1437173A) — 2 doses of HZ/su vaccine were administered intramuscularly according to a 0,2 months vaccination schedule, at Day 1 and Month 2.
  Arms: HZ/su Group
Drug: Placebo — 2 doses of Placebo were administered intramuscularly according to a 0,2 months vaccination schedule, at Day 1 and Month 2.
  Arms: Placebo Group

SUMMARY:
The purpose of this study was to assess the safety and immunogenicity of GSK Biologicals' HZ/su vaccine when given on a two-dose schedule to adults aged 50 years and above who had a previous episode of Herpes Zoster (HZ).

ELIGIBILITY:
Inclusion Criteria:

* Subjects and/or subject's LAR(s) who, in the opinion of the investigator, can and will comply with the requirements of the protocol
* Written informed consent obtained from the subject/subject's LAR(s) prior to performance of any study specific procedure.
* A male or female ≥ 50 YOA at the time of the first vaccination.
* Subjects with a history of HZ. Confirmation of the prior HZ diagnosis can be done by one of the following three methods:

  * Clinically diagnosed HZ:

OR Laboratory diagnosed HZ: OR

* HZ diagnosed by an adjudication committee: Female subjects of non-childbearing potential may be enrolled in the study.
* Non-childbearing potential is defined as current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy, bilateral salpingectomy or post-menopause.

  • Female subjects of childbearing potential may be enrolled in the study if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Subjects who at time of study entry or during the maximum period of anticipated study participation are/will become part of the population recommended to receive a zoster vaccine per existing local or national immunization practices will be excluded from study participation.
* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the first dose of study vaccine, or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Onset of HZ in the past 6 months or any ongoing symptoms from a prior HZ episode.
* Chronic antiviral use for HZ prophylaxis.
* History of >1 prior episode of HZ.
* A history of disseminated HZ, cutaneous or associated with visceral disease or associated with neurologic disease caused by VZV infection.
* Use or anticipated use of immunosuppressants or immune-modifying drugs during the period starting six months prior to study start and during the whole study period. This includes chronic administration of corticosteroids, long-acting immune-modifying agents or immunosuppressive/cytotoxic therapy
* Administration or planned administration of a vaccine not foreseen by the study protocol within the period starting 30 days before the first dose of study vaccine and ending 30 days after the last dose of study vaccine. However, licensed pneumococcal vaccines and non-replicating vaccines may be administered up until 8 days prior to dose 1 and/or dose 2 and/or at least 14 days after any dose of study vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product
* Previous vaccination against VZV or HZ.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Acute disease and/or fever at the time of enrolment.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions in the period up to 2 months after completion of the vaccination series.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1430 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Russia (3):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Gatchina
  - GSK Investigational Site, Moscow

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

REFERENCES:
- [Background] Jegede B, Zhou Y, Hawksworth H, Hui DSC, Montenegro Guerra N, Poder A, Ramon JM, Valimaa H, Villanueva-Quintero GD, Mwakingwe-Omari A; Z-062 study group. Herpes zoster recurrence, and safety and immunogenicity of the recombinant zoster vaccine in adults aged >/=50 years with a history of herpes zoster: A phase 3, randomized controlled trial. J Infect. 2025 Sep;91(3):106573. doi: 10.1016/j.jinf.2025.106573. Epub 2025 Aug 6. PMID 40780591
- [Derived] de Oliveira Gomes J, Gagliardi AM, Andriolo BN, Torloni MR, Andriolo RB, Puga MEDS, Canteiro Cruz E. Vaccines for preventing herpes zoster in older adults. Cochrane Database Syst Rev. 2023 Oct 2;10(10):CD008858. doi: 10.1002/14651858.CD008858.pub5. PMID 37781954

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 46 centers in 8 countries (Estonia, Finland, Hong Kong, Mexico, Panama, Russian Federation, Spain and United Kingdom).
Pre-assignment Details: A total of 1430 participants were enrolled into the study, of which 1426 participants received at least 1 dose of study treatment/vaccine (HZ/su or placebo) and were included in the Exposed Set.
Period: Overall Study
Arm/Group | HZ/su Group | Placebo Group
Started | 714 | 712
Completed | 646 | 640
Not Completed | 68 | 72
Not completed — Adverse Event | 15 | 10
Not completed — Lost to Follow-up | 8 | 8
Not completed — Protocol Violation | 5 | 4
Not completed — Withdrawal by Subject | 21 | 27
Not completed — Non-emergency unblinding/Non-compliance | 15 | 18
Not completed — Migrated/moved from the study area | 3 | 5
Not completed — Suspected HZ episode | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HZ/su Group | Placebo Group | Total
Number analyzed (Participants) | 714 | 712 | 1426
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (8.5) | 64.1 (8.8) | 64.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 430 | 434 | 864
  Male | 284 | 278 | 562
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 80 | 77 | 157
  Not Hispanic or Latino | 634 | 635 | 1269
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate of Confirmed Herpes Zoster (HZ) Cases
Description: A suspected case of HZ is defined as a new unilateral rash accompanied by pain (broadly defined to include allodynia, pruritus or other sensations) and no alternative diagnosis. A suspected case of HZ was confirmed by an algorithm that included Polymerase Chain Reaction (PCR) and the HZ Ascertainment Committee (HZAC) determination. The incidence rate (n/T) of confirmed HZ cases, expressed in terms of 1000 person-years rate, was calculated as the number of participants reporting at least one confirmed HZ case (n) in a group, over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 1000.
Time Frame: From 30 days post-second vaccination (Month 3) until study end (duration of approximately 2 years to 4 years and 5 months)
Population: The analysis was performed on the modified Exposed Set (mES), which excluded participants from the Exposed Set who were not administered 2 doses of the study treatment per protocol, or who developed a confirmed case of HZ prior to 30 days after the second vaccination.
Measure: Number; unit: Cases per 1000 person-years
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 668 | 682
Cases per 1000 person-years | 0.0 | 4.1
Statistical Analysis 1: Comparison: HZ/su Group vs Placebo Group; To demonstrate the non-inferiority of HZ/su vaccine compared to placebo in terms of incidence of HZ recurrence from 30 days post-second vaccination (Month 3) until study end (duration of approximately 2 years to 4 years and 5 months); Test type: Non-Inferiority — The non-inferiority was to be demonstrated if the upper limit (UL) of the 95% confidence interval (CI) of the ratio of the incidence of HZ recurrence between HZ/su group and Placebo group was below (<) 5; Poisson; Incidence Rate Ratio (IRR) = 0.00, 95% CI 2-sided [0.00 to 0.46] — IRR = incidence rate of HZ recurrence in HZ/su group divided by the incidence rate of HZ recurrence in Placebo group. Poisson method was used to adjust for differences in follow-up time across individuals

2. Secondary Outcome: Incidence Rate of Confirmed HZ Cases
Description: A suspected case of HZ is defined as a new unilateral rash accompanied by pain (broadly defined to include allodynia, pruritus or other sensations) and no alternative diagnosis. A suspected case of HZ was confirmed by an algorithm that included PCR and the HZAC determination. The incidence rate (n/T) of confirmed HZ cases, expressed in terms of 1000 person-years rate, was calculated as the number of participants reporting at least one confirmed HZ case (n) in a group, over the sum of follow-up period expressed in years (T) in the same group, and multiplied by 1000.
Time Frame: From first vaccination (Day 1) until study end (duration of approximately 2 years to 4 years and 5 months)
Population: The analysis was performed on the Exposed Set, which included all participants with at least one dose of the study treatment administered.
Measure: Number; unit: Cases per 1000 person-years
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 714 | 712
Cases per 1000 person-years | 0.0 | 3.6

3. Secondary Outcome: Number of Participants With Any and Grade 3 Solicited Administration Site Events
Description: Assessed solicited administration site events included erythema, pain, pruritus and swelling at the injection site. Any = occurrence of the event regardless of intensity grade. Grade 3 pain = significant pain at rest, which prevented normal, everyday activities. Grade 3 erythema, swelling = erythema, swelling with a surface diameter greater than (>) 100 millimeters (mm). Grade 3 pruritus = itchy sensation that prevented normal, everyday activities.
Time Frame: Within 7 days after each vaccination (occurring at Day 1 and Month 2)
Population: The analysis was performed on the Exposed Set, which included all participants with at least one dose of the study treatment administered and with the solicited administration site events diary card data available after the corresponding vaccination for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 697 | 697
Participants
  Any Erythema, post-vaccination at Day 1 | 164 | 5
  Grade 3 Erythema, post-vaccination at Day 1 | 8 | 0
  Any Pain, post-vaccination at Day 1 | 562 | 61
  Grade 3 Pain, post-vaccination at Day 1 | 49 | 2
  Any Pruritus, post-vaccination at Day 1 | 148 | 24
  Grade 3 Pruritus, post-vaccination at Day 1 | 4 | 0
  Any Swelling, post-vaccination at Day 1 | 91 | 1
  Grade 3 Swelling, post-vaccination at Day 1 | 3 | 0
  Any Erythema, post-vaccination at Month 2: number analyzed (Participants) | 669 | 682
  Any Erythema, post-vaccination at Month 2 | 164 | 0
  Grade 3 Erythema, post-vaccination at Month 2: number analyzed (Participants) | 669 | 682
  Grade 3 Erythema, post-vaccination at Month 2 | 14 | 0
  Any Pain, post-vaccination at Month 2: number analyzed (Participants) | 669 | 682
  Any Pain, post-vaccination at Month 2 | 503 | 48
  Grade 3 Pain, post-vaccination at Month 2: number analyzed (Participants) | 669 | 682
  Grade 3 Pain, post-vaccination at Month 2 | 48 | 0
  Any Pruritus, post-vaccination at Month 2: number analyzed (Participants) | 669 | 682
  Any Pruritus, post-vaccination at Month 2 | 142 | 10
  Grade 3 Pruritus, post-vaccination at Month 2: number analyzed (Participants) | 669 | 682
  Grade 3 Pruritus, post-vaccination at Month 2 | 7 | 0
  Any Swelling, post-vaccination at Month 2: number analyzed (Participants) | 669 | 682
  Any Swelling, post-vaccination at Month 2 | 82 | 1
  Grade 3 Swelling, post-vaccination at Month 2: number analyzed (Participants) | 669 | 682
  Grade 3 Swelling, post-vaccination at Month 2 | 3 | 0

4. Secondary Outcome: Duration in Days of Solicited Administration Site Events
Description: Duration is the number of days in which a participant experienced the symptom within the 7-day solicited follow-up period. Assessed solicited administration site events included erythema, pain, pruritus and swelling at the injection site.
Time Frame: Within 7 days after each vaccination (occurring at Day 1 and Month 2)
Population: The analysis was performed on the Exposed Set, which included all participants with at least one dose of the study treatment administered, with solicited diary data available after the corresponding vaccination and who experienced the specified solicited administration site event within 7 days following the respective study treatment dose. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 562 | 61
Days
  Erythema, post-vaccination at Day 1: number analyzed (Participants) | 164 | 5
  Erythema, post-vaccination at Day 1 | 3.0 [2.0 to 5.0] | 3.0 [2.0 to 4.0]
  Pain, post-vaccination at Day 1 | 3.0 [2.0 to 4.0] | 1.0 [1.0 to 2.0]
  Pruritus, post-vaccination at Day 1: number analyzed (Participants) | 148 | 24
  Pruritus, post-vaccination at Day 1 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Swelling, post-vaccination at Day 1: number analyzed (Participants) | 91 | 1
  Swelling, post-vaccination at Day 1 | 3.0 [1.0 to 4.0] | 2.0 [2.0 to 2.0]
  Erythema, post-vaccination at Month 2: number analyzed (Participants) | 164 | 0
  Erythema, post-vaccination at Month 2 | 3.0 [2.0 to 5.0] |
  Pain, post-vaccination at Month 2: number analyzed (Participants) | 503 | 48
  Pain, post-vaccination at Month 2 | 3.0 [2.0 to 4.0] | 1.0 [1.0 to 2.0]
  Pruritus, post-vaccination at Month 2: number analyzed (Participants) | 142 | 10
  Pruritus, post-vaccination at Month 2 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Swelling, post-vaccination at Month 2: number analyzed (Participants) | 82 | 1
  Swelling, post-vaccination at Month 2 | 3.0 [2.0 to 4.0] | 6.0 [6.0 to 6.0]

5. Secondary Outcome: Number of Participants With Any, Grade 3 and Related Solicited Systemic Events
Description: Assessed solicited systemic events included fatigue, fever (defined as axillary temperature greater than or equal to (>=) 38.0°C/100.4°F), gastrointestinal symptoms, headache, malaise, myalgia, and shivering. Any = occurrence of the event regardless of intensity grade or relation to the study vaccination. Grade 3 = event that prevented normal, everyday activities. Grade 3 fever = axillary temperature higher than (>) 39.0°C/102.2°F. Related = event assessed by the investigator as related to the study vaccination.
Time Frame: Within 7 days after each vaccination (occurring at Day 1 and Month 2)
Population: The analysis was performed on the Exposed Set, which included all participants with at least one dose of the study treatment administered and with the solicited systemic events diary card data available after the corresponding vaccination for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 698 | 697
Participants
  Any Fatigue, post-vaccination at Day 1 | 329 | 146
  Grade 3 Fatigue, post-vaccination at Day 1 | 42 | 10
  Related Fatigue, post-vaccination at Day 1 | 292 | 105
  Any Fever, post-vaccination at Day 1 | 26 | 4
  Grade 3 Fever, post-vaccination at Day 1 | 1 | 0
  Related Fever, post-vaccination at Day 1 | 26 | 4
  Any Gastrointestinal symptoms, post-vaccination at Day 1 | 103 | 79
  Grade 3 Gastrointestinal symptoms, post-vaccination at Day 1 | 8 | 4
  Related Gastrointestinal symptoms, post-vaccination at Day 1 | 84 | 54
  Any Headache, post-vaccination at Day 1 | 266 | 136
  Grade 3 Headache, post-vaccination at Day 1 | 21 | 11
  Related Headache, post-vaccination at Day 1 | 224 | 90
  Any Malaise, post-vaccination at Day 1 | 260 | 70
  Grade 3 Malaise, post-vaccination at Day 1 | 30 | 9
  Related Malaise, post-vaccination at Day 1 | 231 | 52
  Any Myalgia, post-vaccination at Day 1 | 262 | 65
  Grade 3 Myalgia, post-vaccination at Day 1 | 17 | 8
  Related Myalgia, post-vaccination at Day 1 | 240 | 45
  Any Shivering, post-vaccination at Day 1 | 185 | 43
  Grade 3 Shivering, post-vaccination at Day 1 | 16 | 0
  Related Shivering, post-vaccination at Day 1 | 174 | 36
  Any Fatigue, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Any Fatigue, post-vaccination at Month 2 | 364 | 115
  Grade 3 Fatigue, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Grade 3 Fatigue, post-vaccination at Month 2 | 59 | 10
  Related Fatigue, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Related Fatigue, post-vaccination at Month 2 | 327 | 85
  Any Fever, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Any Fever, post-vaccination at Month 2 | 66 | 5
  Grade 3 Fever, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Grade 3 Fever, post-vaccination at Month 2 | 4 | 1
  Related Fever, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Related Fever, post-vaccination at Month 2 | 63 | 3
  Any Gastrointestinal symptoms, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Any Gastrointestinal symptoms, post-vaccination at Month 2 | 118 | 54
  Grade 3 Gastrointestinal symptoms, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Grade 3 Gastrointestinal symptoms, post-vaccination at Month 2 | 11 | 4
  Related Gastrointestinal symptoms, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Related Gastrointestinal symptoms, post-vaccination at Month 2 | 102 | 37
  Any Headache, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Any Headache, post-vaccination at Month 2 | 290 | 113
  Grade 3 Headache, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Grade 3 Headache, post-vaccination at Month 2 | 30 | 6
  Related Headache, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Related Headache, post-vaccination at Month 2 | 256 | 73
  Any Malaise, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Any Malaise, post-vaccination at Month 2 | 321 | 69
  Grade 3 Malaise, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Grade 3 Malaise, post-vaccination at Month 2 | 45 | 7
  Related Malaise, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Related Malaise, post-vaccination at Month 2 | 290 | 50
  Any Myalgia, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Any Myalgia, post-vaccination at Month 2 | 294 | 54
  Grade 3 Myalgia, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Grade 3 Myalgia, post-vaccination at Month 2 | 41 | 2
  Related Myalgia, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Related Myalgia, post-vaccination at Month 2 | 269 | 40
  Any Shivering, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Any Shivering, post-vaccination at Month 2 | 253 | 32
  Grade 3 Shivering, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Grade 3 Shivering, post-vaccination at Month 2 | 37 | 2
  Related Shivering, post-vaccination at Month 2: number analyzed (Participants) | 671 | 680
  Related Shivering, post-vaccination at Month 2 | 234 | 28

6. Secondary Outcome: Duration in Days of Solicited Systemic Events
Description: Duration is the number of days in which a participant experienced the symptom within the 7-day solicited follow-up period. Assessed solicited systemic events included fatigue, fever (defined as axillary temperature >=38.0°C/100.4°F), gastrointestinal symptoms, headache, malaise, myalgia and shivering.
Time Frame: Within 7 days after each vaccination (occurring at Day 1 and Month 2)
Population: The analysis was performed on the Exposed Set, which included all participants with at least one dose of the study treatment administered, with solicited diary data available after the corresponding vaccination and who experienced the specified solicited systemic event within 7 days following the respective study treatment dose. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 364 | 146
Days
  Fatigue, post-vaccination at Day 1: number analyzed (Participants) | 329 | 146
  Fatigue, post-vaccination at Day 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Fever, post-vaccination at Day 1: number analyzed (Participants) | 26 | 4
  Fever, post-vaccination at Day 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Gastrointestinal symptoms, post-vaccination at Day 1: number analyzed (Participants) | 103 | 79
  Gastrointestinal symptoms, post-vaccination at Day 1 | 1.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0]
  Headache, post-vaccination at Day 1: number analyzed (Participants) | 266 | 136
  Headache, post-vaccination at Day 1 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 3.0]
  Malaise, post-vaccination at Day 1: number analyzed (Participants) | 260 | 70
  Malaise, post-vaccination at Day 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Myalgia, post-vaccination at Day 1: number analyzed (Participants) | 262 | 65
  Myalgia, post-vaccination at Day 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Shivering, post-vaccination at Day 1: number analyzed (Participants) | 185 | 43
  Shivering, post-vaccination at Day 1 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Fatigue, post-vaccination at Month 2: number analyzed (Participants) | 364 | 115
  Fatigue, post-vaccination at Month 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Fever, post-vaccination at Month 2: number analyzed (Participants) | 66 | 5
  Fever, post-vaccination at Month 2 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Gastrointestinal symptoms, post-vaccination at Month 2: number analyzed (Participants) | 118 | 54
  Gastrointestinal symptoms, post-vaccination at Month 2 | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Headache, post-vaccination at Month 2: number analyzed (Participants) | 290 | 113
  Headache, post-vaccination at Month 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0]
  Malaise, post-vaccination at Month 2: number analyzed (Participants) | 321 | 69
  Malaise, post-vaccination at Month 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0]
  Myalgia, post-vaccination at Month 2: number analyzed (Participants) | 294 | 54
  Myalgia, post-vaccination at Month 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 5.0]
  Shivering, post-vaccination at Month 2: number analyzed (Participants) | 253 | 32
  Shivering, post-vaccination at Month 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0]

7. Secondary Outcome: Number of Participants With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE is defined as any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event. Any = occurrence the event regardless of intensity grade or relation to the study vaccination. Grade 3 = event that prevented normal, everyday activities. Related = event assessed by the investigator as related to the study vaccination.
Time Frame: Within 30 days after each vaccination (occurring at Day 1 and Month 2)
Population: The analysis was performed on the Exposed Set, which included all participants with at least one dose of the study treatment administered and for whom unsolicited AEs data were available for the specified duration after each vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 714 | 712
Participants
  Any Unsolicited AEs, post-vaccination at Day 1 | 118 | 104
  Grade 3 Unsolicited AEs, post-vaccination at Day 1 | 12 | 10
  Related Unsolicited AEs, post-vaccination at Day 1 | 32 | 18
  Any Unsolicited AEs, post-vaccination at Month 2: number analyzed (Participants) | 675 | 686
  Any Unsolicited AEs, post-vaccination at Month 2 | 120 | 116
  Grade 3 Unsolicited AEs, post-vaccination at Month 2: number analyzed (Participants) | 675 | 686
  Grade 3 Unsolicited AEs, post-vaccination at Month 2 | 13 | 6
  Related Unsolicited AEs, post-vaccination at Month 2: number analyzed (Participants) | 675 | 686
  Related Unsolicited AEs, post-vaccination at Month 2 | 33 | 7

8. Secondary Outcome: Number of Participants With Any and Related Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study participant. Any = occurrence of the SAE regardless of intensity grade or relation to the study vaccination. Related = SAE assessed by the investigator as related to the study vaccination.
Time Frame: From first vaccination (Day 1) to 30 days post-last vaccination (last vaccination administered at Day 1 for participants who received only 1 dose and at Month 2 for participants who received 2 doses)
Population: The analysis was performed on the Exposed Set, which included all participants with at least one dose of the study treatment administered and for whom SAEs data were available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 714 | 712
Participants
  Any SAEs | 11 | 11
  Related SAEs | 0 | 0

9. Secondary Outcome: Number of Participants With Any and Related Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs are defined as a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Any = occurrence of the pIMD regardless of intensity grade or relation to the study vaccination. Related = pIMD assessed by the investigator as related to the study vaccination.
Time Frame: as for outcome 8
Population: The analysis was performed on the Exposed Set, which included all participants with at least one dose of the study treatment administered and for whom pIMDs data were available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 714 | 712
Participants
  Any pIMDs | 2 | 2
  Related pIMDs | 0 | 1

10. Secondary Outcome: Number of Participants With Any and Related SAEs
Description: as for outcome 8
Time Frame: From 30 days post-last vaccination until 1 year post-last vaccination (last vaccination administered at Day 1 for participants who received only 1 dose and at Month 2 for participants who received 2 doses)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 714 | 712
Participants
  Any SAEs | 35 | 22
  Related SAEs | 0 | 0

11. Secondary Outcome: Number of Participants With Any and Related pIMDs
Description: as for outcome 9
Time Frame: as for outcome 10
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 714 | 712
Participants
  Any pIMDs | 2 | 5
  Related pIMDs | 0 | 0

12. Secondary Outcome: Number of Participants With SAEs Related to Investigational Vaccine, Related to Study Participation or to GSK Concomitant Medication/Vaccine
Description: An SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study participant. Any SAEs related to the investigational vaccine or related to study participation or to a GSK concomitant medication/vaccine as assessed by the investigator are reported.
Time Frame: From first vaccination (Day 1) until study end (duration of approximately 2 years to 4 years and 5 months)
Population: The analysis was performed on the Exposed Set, which included all participants with at least one dose of the study treatment administered and for whom SAEs related to investigational vaccine/study participation/GSK concomitant medication/vaccine data were available for the specified duration.
Measure: Count of Participants; unit: Participants
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 714 | 712
Participants | 1 | 1

13. Secondary Outcome: Percentage of Participants With Vaccine Response for Anti-glycoprotein E (Anti-gE) Antibodies as Determined by Enzyme Linked Immunosorbent Assay (ELISA)
Description: Vaccine response for anti-gE antibodies is defined as:
  * For initially seronegative participants, anti-gE antibody concentration at post-vaccination >= 4-fold the cut-off value for anti-gE [97 international units per liter (IU/L)].
  * For initially seropositive participants, anti-gE antibody concentration at post-vaccination >= 4-fold the pre-vaccination anti-gE antibody concentration.
Time Frame: At Month 2 and Month 3
Population: The analysis was performed on the Adapted Per Protocol Set for immunogenicity, which included all evaluable participants from the Exposed Set who met all eligibility criteria, received 2 doses of the HZ/su vaccine/placebo according to their random assignment, did not receive forbidden medications, had no intercurrent medical condition complied with the vaccination and blood sample schedules and for whom results were available for the specified analysis at the specified time points.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 593 | 592
Percentage of participants
  At Month 2 | 85.8 [82.8 to 88.5] | 0.2 [0.0 to 0.9]
  At Month 3: number analyzed (Participants) | 531 | 521
  At Month 3 | 95.3 [93.1 to 96.9] | 0.2 [0.0 to 1.1]

14. Secondary Outcome: Anti-gE Antibody Concentrations Expressed as Geometric Mean Concentrations (GMCs) as Determined by ELISA
Description: Anti-gE antibody concentrations were determined by ELISA and expressed as GMCs in IU/L.
Time Frame: At Day 1, Month 2 and Month 3
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: IU/L
Arm/Group | HZ/su Group | Placebo Group
Number analyzed (Participants) | 664 | 658
IU/L
  At Day 1 | 2151.30 [2004.22 to 2309.17] | 2087.14 [1942.47 to 2242.58]
  At Month 2: number analyzed (Participants) | 596 | 599
  At Month 2 | 24346.52 [22840.59 to 25951.74] | 1850.11 [1725.86 to 1983.30]
  At Month 3: number analyzed (Participants) | 534 | 526
  At Month 3 | 49175.78 [46500.40 to 52005.09] | 1849.08 [1718.02 to 1990.13]

ADVERSE EVENTS:
Time Frame: Solicited AEs: within 7 days after any vaccination. Unsolicited AEs: within 30 days after any vaccination. All-cause mortality & SAEs: from first vaccination (Day 1) until study end (duration of approximately 2 years to 4 years and 5 months). pIMDs: from first vaccination (Day 1) until 1 year post-last vaccination (last vaccination administered at Day 1 for participants who received only 1 dose and at Month 2 for participants who received 2 doses).
Description: All events presented in the All-cause mortality, Serious Adverse Events and Other (not including Serious) Adverse Events modules are reported for the Exposed Set population during the specified time frames.
  All SAEs regardless of relation to study vaccine/study participation/GSK concomitant medication/vaccination are reported in the Serious Adverse Events module.
Arm/Group | HZ/su Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 12/714 | 8/712
Serious Adverse Events (participants affected / at risk) | 56/714 | 43/712
Other Adverse Events (participants affected / at risk) | 665/714 | 414/712
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HZ/su Group (N=714) | Placebo Group (N=712)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (3)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary dilatation (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 4 (4) | 5 (5)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Neurosyphilis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Costal cartilage fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leiomyosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Splenic marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HZ/su Group (N=714) | Placebo Group (N=712)
Administration site pain (General disorders) | 611 (1065) | 94 (109)
Fatigue (General disorders) | 457 (695) | 199 (262)
Malaise (General disorders) | 396 (584) | 112 (139)
Chills (General disorders) | 330 (440) | 64 (76)
Administration site erythema (General disorders) | 238 (328) | 5 (5)
Administration site swelling (General disorders) | 133 (173) | 2 (2)
Pyrexia (General disorders) | 88 (94) | 10 (10)
Injection site bruising (General disorders) | 2 (2) | 1 (1)
Asthenia (General disorders) | 2 (2) | 0 (0)
Feeling hot (General disorders) | 1 (3) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 2 (2)
Injection site rash (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Swelling (General disorders) | 2 (2) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1)
Illness (General disorders) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0)
Injection site hypoaesthesia (General disorders) | 0 (0) | 1 (1)
Injection site joint pain (General disorders) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 1 (1) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Temperature regulation disorder (General disorders) | 1 (1) | 0 (0)
Vaccination site movement impairment (General disorders) | 1 (1) | 0 (0)
Vaccination site pain (General disorders) | 1 (1) | 0 (0)
Vaccination site scar (General disorders) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 384 (573) | 201 (270)
Dizziness (Nervous system disorders) | 5 (5) | 3 (3)
Paraesthesia (Nervous system disorders) | 3 (4) | 4 (4)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 389 (560) | 97 (122)
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (24) | 8 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (6) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 5 (5)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 179 (221) | 117 (134)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 2 (2) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hyperchlorhydria (Gastrointestinal disorders) | 0 (0) | 1 (2)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 228 (297) | 33 (41)
Erythema (Skin and subcutaneous tissue disorders) | 10 (11) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 18 (19) | 16 (19)
COVID-19 (Infections and infestations) | 8 (8) | 8 (8)
Oral herpes (Infections and infestations) | 9 (9) | 6 (6)
Urinary tract infection (Infections and infestations) | 3 (3) | 5 (5)
Influenza (Infections and infestations) | 4 (4) | 3 (3)
Sinusitis (Infections and infestations) | 2 (3) | 3 (3)
Conjunctivitis (Infections and infestations) | 1 (1) | 3 (3)
Otitis externa (Infections and infestations) | 2 (2) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3)
Acute sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 2 (2) | 1 (1)
Herpes simplex (Infections and infestations) | 3 (3) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Suspected COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Tinea pedis (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Bartholinitis (Infections and infestations) | 1 (1) | 0 (0)
Borrelia infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Furuncle (Infections and infestations) | 0 (0) | 1 (1)
Genital herpes (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Pustule (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in throat (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (3) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Middle insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Persistent depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Terminal insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 3 (3)
Hypertensive crisis (Vascular disorders) | 2 (2) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 2 (2)
Vitreous detachment (Eye disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Erythema of eyelid (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0)
Iridocyclitis (Eye disorders) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 1 (1) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 3 (3)
Bladder discomfort (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 1 (2)
Hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital erythema (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic lesion (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0)
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/51/NCT04091451/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT04091451/SAP_001.pdf